CLINICAL TRIAL: NCT00928109
Title: Innovative Trial for the Treatment of Anorexia Nervosa in Late Adolescence and Adulthood
Brief Title: UCAN: Uniting Couples in the Treatment of Anorexia Nervosa
Acronym: UCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07-1429; R01MH082732-01 (NIH)
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Anorexia Nervosa
Keywords: eating disorders; couples therapy
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavioral Couples Therapy (CBCT) (Experimental): CBCT is a 20-week program consisting of 1-hour sessions between a couple and a therapist. In this program, couples learn about ways to communicate about their relationship in the context of experiencing anorexia nervosa. CBCT focuses on couple-specific skills such as communication and targets relationship domains such as exercise, body image and sexuality, eating together as a couple, and broader relationship concerns outside of anorexia nervosa.
  Interventions: Behavioral: CBCT
- Family Supportive Therapy (Active Comparator): Couples meet once a week for an hour for a period of 20 weeks for couples therapy. Family Supportive Therapy is not manualized and is the standard form of care at the UNC Eating Disorders Program
  Interventions: Behavioral: Family Supportive Therapy

INTERVENTIONS:
Behavioral: CBCT — Cognitive Behavioral Couples Therapy - weekly manualized couples therapy
  Other Names: UCAN
  Arms: Cognitive Behavioral Couples Therapy (CBCT)
Behavioral: Family Supportive Therapy — Couples meet once a week for an hour for a period of 20 weeks for couples therapy. Family Supportive Therapy is not manualized and is the standard form of care at the UNC Eating Disorders Program
  Other Names: Eating Disorder Treatment as Usual
  Arms: Family Supportive Therapy

SUMMARY:
UCAN is a research program funded by the National Institute of Mental Health and is part of the UNC Eating Disorders Program. UCAN aims to help couples work together in the treatment of anorexia nervosa. Couples participate in UCAN over a period of six months and return for follow-up treatment three months after the end of the original six-month period. Patients receive weekly individual therapy, monthly psychiatry consultations, monthly dietary consultations in addition to being randomized to one of two types of weekly couples therapy. Participation in UCAN can help participants gain new confidence in facing anorexia as a team and can help us understand how best to involve partners in the treatment of eating disorders.

DETAILED DESCRIPTION:
Patients receive comprehensive eating disorder treatment at the UNC Eating Disorders Outpatient Program in addition to couples therapy. Eligibility: Participants may be eligible if they are 18 or older, have anorexia nervosa and are currently living with a partner with whom they have been in a committed relationship for at least a year. The partner must also be willing to enter treatment.

ELIGIBILITY:
Inclusion Criteria:

* Anorexia Nervosa,
* 18 years or older,
* BMI 16 or higher,
* In a committed relationship with a partner for 1 year or longer and currently living together.

Exclusion Criteria:

* Alcohol or drug dependence in past year,
* Current significant suicidal ideation,
* Developmental disability that would impair the ability of the participant to benefit from the intervention,
* Psychosis,
* BMI less than 16.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Eating disorder behavior | 9 months

SECONDARY OUTCOMES:
Couple Satisfaction | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia M Bulik, PhD, Principal Investigator — UNC Chapel Hill Department of Psychiatry; Donald Baucom, PhD, Principal Investigator — UNC Chapel Hill Department of Psychology
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States